CLINICAL TRIAL: NCT05527782
Title: A Phase II Study of Efficacy and Safety of Induction Modified TPF (mTPF) Followed by Concurrent Chemoradiotherapy (CCRT) in Locally Advanced Squamous Cell Carcinoma of the Head and Neck (LASCCHN)
Brief Title: Induction Modified TPF Followed by Concurrent Chemoradiotherapy in Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitario Doctor Peset (Other)
Responsible Party: Principal Investigator, Sebastian Ochenduszko, Attending Physician, Hospital Universitario Doctor Peset
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUDP-CyC-01/2022
Record Dates: First submitted 2022-08-31; First posted 2022-09-06 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Locally Advanced Head and Neck Squamous Cell Carcinoma
Keywords: head and neck cancer; induction chemotherapy; modified TPF; concurrent chemoradiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- induction mTPF (Experimental): 1. 4 CYCLES OF INDUCTION mTPF: Docetaxel 40 mg/m2 iv day 1, Cisplatin 40 mg/m2 iv day 1, Leucovorin 400 mg/m2 iv followed by Fluorouracil (5FU) bolus 400 mg/m2 iv day 1, 5FU 1000 mg/m2 iv day 1-2, q2w. Primary neutropenic fever prophylaxis with GCSFs x 3 days
  2. CONCURRENT CHEMORADIOTHERAPY WITH 2 CYCLES OF CISPLATIN 100mg/m2 iv q3w
  Interventions: Drug: modified TPF; Other: Quality of life assessment (QoL)

INTERVENTIONS:
Drug: modified TPF — modified TPF: modified docetaxel-cisplatin-fluorouracil followed by concurrent chemoradiotherapy
Other: Quality of life assessment (QoL) — Quality of life assessment with questionnaires: EORTC QLQ-C30 and QLQ H&N-35

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of induction mTPF chemotherapy followed by concurrent chemoradiotherapy for locally advanced squamous cell carcinoma of the head and neck cancer

DETAILED DESCRIPTION:
The prognosis of patients with locally advanced squamous cell carcinoma of the head and neck (LASCCHN) is poor, therefore continuous research effort is being made in order to improve treatment efficacy. Standard treatment consists of concurrent chemoradiotherapy (CCRT) with cisplatin. In spite of many clinical trials and meta-analyses, the improvement of patient outcomes with the use of induction chemotherapy (IC) hasn´t been clearly demonstrated, partially due to the high toxicity of the standard TPF (docetaxel+cisplatin+fluorouracil) regimen used most frequently in this setting. Therefore, the aim of this study is to evaluate the outcomes of patients with LASCCHN treated with a less toxic induction mTPF regimen followed by CCRT.

The study will include patients with LASCCHN who - by the decision of the multidisciplinary team - have been assigned treatment with IC followed by CCRT. After being informed about the study objectives and potential risks, all patients giving written informed consent and meeting all the eligibility criteria will start the treatment. According to the study protocol, participants will receive 4 cycles of induction mTPF regimen repeated every 2 weeks followed by computed tomography (CT) response evaluation. 3-6 weeks after having completed the last cycle of mTPF, patients without disease progression will start CCRT with 2 cycles of cisplatin every 3 weeks. Twelve weeks after radiotherapy termination, a PET-CT scan will be performed in order to evaluate the treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* patients with locally advanced squamous cell carcinoma of the head and neck (LASCCHN): oral cavity, oropharynx, larynx, hypopharynx, and unknown primary
* stage cT4 and/or cN2-N3, with no distant metastases (M0).
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-2
* initial clinical staging evaluated in:

  1. CT scan or MRI of the neck and CT scan of the chest or
  2. FDG18 PET TC

Exclusion Criteria:

* patients with p16 positive oropharyngeal carcinoma cT0-T3 N2 M0 (stage II), unless extranodal tumor extension
* contraindications for cisplatin administration: renal insufficiency (eGFR < 55ml/min), hearing loss, peripheral neuropathy
* dysphagia G>2 with no percutaneous gastrostomy
* the presence of distant metastasis (M1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | 12 weeks after radiotherapy termination
  percentage of partial and complete response rates (RR)

SECONDARY OUTCOMES:
24 month progression free survival (PFS) | 2 years
  PFS at 24 months after treatment initiation
24 month overall survival (OS) | 2 years
  OS at 24 months after treatment initiation
toxicity of induction mTPF | up to 10 weeks
  percentages of patients with adverse effects during induction mTPF
toxicity of concurrent chemoradiotherapy (CCRT) | through study completion, an average of 2 years
  percentages of patients with adverse effects during CCRT
EORTC Core Quality of Life questionnaire (EORTC QLQ-C30) | 9 months
  measurement of patients' physical, psychological and social functions
EORTC Head and Neck Cancer specific module (EORTC QLQ-H&N35) | 9 months
  assessment the HR-QoL specific for head-and-neck cancer patients

OTHER OUTCOMES:
treatment compliance according to the protocol | 2 years
  percentage of patients that have completed the sequence of induction mTPF followed by CCRT
treatment dose modifications and delays | 2 years
  percentage of patients that have required dose reductions and/or delays in the administration of induction mTPF

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Marina Baixa, Villajoyosa, Alicante
  - Hospital Comarcal Francesc De Borja, Gandia, Valencia
  - Hospital Universitario Doctor Peset, Valencia

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Forastiere AA, Zhang Q, Weber RS, Maor MH, Goepfert H, Pajak TF, Morrison W, Glisson B, Trotti A, Ridge JA, Thorstad W, Wagner H, Ensley JF, Cooper JS. Long-term results of RTOG 91-11: a comparison of three nonsurgical treatment strategies to preserve the larynx in patients with locally advanced larynx cancer. J Clin Oncol. 2013 Mar 1;31(7):845-52. doi: 10.1200/JCO.2012.43.6097. Epub 2012 Nov 26. PMID 23182993
- [Background] Department of Veterans Affairs Laryngeal Cancer Study Group; Wolf GT, Fisher SG, Hong WK, Hillman R, Spaulding M, Laramore GE, Endicott JW, McClatchey K, Henderson WG. Induction chemotherapy plus radiation compared with surgery plus radiation in patients with advanced laryngeal cancer. N Engl J Med. 1991 Jun 13;324(24):1685-90. doi: 10.1056/NEJM199106133242402. PMID 2034244
- [Background] Blanchard P, Baujat B, Holostenco V, Bourredjem A, Baey C, Bourhis J, Pignon JP; MACH-CH Collaborative group. Meta-analysis of chemotherapy in head and neck cancer (MACH-NC): a comprehensive analysis by tumour site. Radiother Oncol. 2011 Jul;100(1):33-40. doi: 10.1016/j.radonc.2011.05.036. Epub 2011 Jun 16. PMID 21684027
- [Background] Posner MR, Hershock DM, Blajman CR, Mickiewicz E, Winquist E, Gorbounova V, Tjulandin S, Shin DM, Cullen K, Ervin TJ, Murphy BA, Raez LE, Cohen RB, Spaulding M, Tishler RB, Roth B, Viroglio Rdel C, Venkatesan V, Romanov I, Agarwala S, Harter KW, Dugan M, Cmelak A, Markoe AM, Read PW, Steinbrenner L, Colevas AD, Norris CM Jr, Haddad RI; TAX 324 Study Group. Cisplatin and fluorouracil alone or with docetaxel in head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1705-15. doi: 10.1056/NEJMoa070956. PMID 17960013
- [Background] Vermorken JB, Remenar E, van Herpen C, Gorlia T, Mesia R, Degardin M, Stewart JS, Jelic S, Betka J, Preiss JH, van den Weyngaert D, Awada A, Cupissol D, Kienzer HR, Rey A, Desaunois I, Bernier J, Lefebvre JL; EORTC 24971/TAX 323 Study Group. Cisplatin, fluorouracil, and docetaxel in unresectable head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1695-704. doi: 10.1056/NEJMoa071028. PMID 17960012
- [Background] Blanchard P, Bourhis J, Lacas B, Posner MR, Vermorken JB, Cruz Hernandez JJ, Bourredjem A, Calais G, Paccagnella A, Hitt R, Pignon JP; Meta-Analysis of Chemotherapy in Head and Neck Cancer, Induction Project, Collaborative Group. Taxane-cisplatin-fluorouracil as induction chemotherapy in locally advanced head and neck cancers: an individual patient data meta-analysis of the meta-analysis of chemotherapy in head and neck cancer group. J Clin Oncol. 2013 Aug 10;31(23):2854-60. doi: 10.1200/JCO.2012.47.7802. Epub 2013 Jul 8. PMID 23835714
- [Background] Haddad R, O'Neill A, Rabinowits G, Tishler R, Khuri F, Adkins D, Clark J, Sarlis N, Lorch J, Beitler JJ, Limaye S, Riley S, Posner M. Induction chemotherapy followed by concurrent chemoradiotherapy (sequential chemoradiotherapy) versus concurrent chemoradiotherapy alone in locally advanced head and neck cancer (PARADIGM): a randomised phase 3 trial. Lancet Oncol. 2013 Mar;14(3):257-64. doi: 10.1016/S1470-2045(13)70011-1. Epub 2013 Feb 13. PMID 23414589
- [Background] Cohen EE, Karrison TG, Kocherginsky M, Mueller J, Egan R, Huang CH, Brockstein BE, Agulnik MB, Mittal BB, Yunus F, Samant S, Raez LE, Mehra R, Kumar P, Ondrey F, Marchand P, Braegas B, Seiwert TY, Villaflor VM, Haraf DJ, Vokes EE. Phase III randomized trial of induction chemotherapy in patients with N2 or N3 locally advanced head and neck cancer. J Clin Oncol. 2014 Sep 1;32(25):2735-43. doi: 10.1200/JCO.2013.54.6309. Epub 2014 Jul 21. PMID 25049329
- [Background] Burgy M, Leblanc J, Borel C. Any place left for induction chemotherapy for locally advanced head and neck squamous cell carcinoma? Anticancer Drugs. 2018 Apr;29(4):287-294. doi: 10.1097/CAD.0000000000000595. PMID 29420335
- [Background] Hitt R, Grau JJ, Lopez-Pousa A, Berrocal A, Garcia-Giron C, Irigoyen A, Sastre J, Martinez-Trufero J, Brandariz Castelo JA, Verger E, Cruz-Hernandez JJ; Spanish Head and Neck Cancer Cooperative Group (TTCC). A randomized phase III trial comparing induction chemotherapy followed by chemoradiotherapy versus chemoradiotherapy alone as treatment of unresectable head and neck cancer. Ann Oncol. 2014 Jan;25(1):216-25. doi: 10.1093/annonc/mdt461. Epub 2013 Nov 19. PMID 24256848
- [Background] Driessen CM, de Boer JP, Gelderblom H, Rasch CR, de Jong MA, Verbist BM, Melchers WJ, Tesselaar ME, van der Graaf WT, Kaanders JH, van Herpen CM. Induction chemotherapy with docetaxel/cisplatin/5-fluorouracil followed by randomization to two cisplatin-based concomitant chemoradiotherapy schedules in patients with locally advanced head and neck cancer (CONDOR study) (Dutch Head and Neck Society 08-01): A randomized phase II study. Eur J Cancer. 2016 Jan;52:77-84. doi: 10.1016/j.ejca.2015.09.024. Epub 2015 Dec 1. PMID 26655558
- [Background] Kim R, Hahn S, Shin J, Ock CY, Kim M, Keam B, Kim TM, Kim DW, Heo DS. The Effect of Induction Chemotherapy Using Docetaxel, Cisplatin, and Fluorouracil on Survival in Locally Advanced Head and Neck Squamous Cell Carcinoma: A Meta-Analysis. Cancer Res Treat. 2016 Jul;48(3):907-16. doi: 10.4143/crt.2015.359. Epub 2015 Nov 17. PMID 26582394
- [Background] Lau A, Li KY, Yang WF, Su YX. Induction chemotherapy for squamous cell carcinomas of the oral cavity: A cumulative meta-analysis. Oral Oncol. 2016 Oct;61:104-14. doi: 10.1016/j.oraloncology.2016.08.022. Epub 2016 Sep 7. PMID 27688112
- [Background] Jerzak KJ, Delos Santos K, Saluja R, Lien K, Lee J, Chan KKW. A network meta-analysis of the sequencing and types of systemic therapies with definitive radiotherapy in locally advanced squamous cell carcinoma of the head and neck (LASCCHN)☆. Oral Oncol. 2017 Aug;71:1-10. doi: 10.1016/j.oraloncology.2017.05.011. Epub 2017 Jun 3. PMID 28688674
- [Background] Ghi MG, Paccagnella A, Ferrari D, Foa P, Alterio D, Codeca C, Nole F, Verri E, Orecchia R, Morelli F, Parisi S, Mastromauro C, Mione CA, Rossetto C, Polsinelli M, Koussis H, Loreggian L, Bonetti A, Campostrini F, Azzarello G, D'Ambrosio C, Bertoni F, Casanova C, Emiliani E, Guaraldi M, Bunkheila F, Bidoli P, Niespolo RM, Gava A, Massa E, Frattegiani A, Valduga F, Pieri G, Cipani T, Da Corte D, Chiappa F, Rulli E; GSTTC (Gruppo di Studio Tumori della Testa e del Collo) Italian Study Group. Induction TPF followed by concomitant treatment versus concomitant treatment alone in locally advanced head and neck cancer. A phase II-III trial. Ann Oncol. 2017 Sep 1;28(9):2206-2212. doi: 10.1093/annonc/mdx299. PMID 28911070
- [Background] Fayette J, Fontaine-Delaruelle C, Ambrun A, Daveau C, Poupart M, Ramade A, Zrounba P, Neidhardt EM, Peron J, Diallo A, Ceruse P. Neoadjuvant modified TPF (docetaxel, cisplatin, fluorouracil) for patients unfit to standard TPF in locally advanced head and neck squamous cell carcinoma: a study of 48 patients. Oncotarget. 2016 Jun 14;7(24):37297-37304. doi: 10.18632/oncotarget.8934. PMID 27119503